CLINICAL TRIAL: NCT00019656
Title: A Phase I Trial of Oral Perifosine With Different Loading Schedules in Patients With Refractory Neoplasms
Brief Title: Perifosine in Treating Patients With Refractory Solid Tumors or Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066960; NCI-99-C-0043; NCI-T98-0065; NCT00001799 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2004-08

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; unspecified adult solid tumor, protocol specific; previously treated myelodysplastic syndromes; de novo myelodysplastic syndromes; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; secondary myelodysplastic syndromes; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; chronic myelomonocytic leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone | interventions — perifosine

INTERVENTIONS:
Drug: perifosine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of perifosine in treating patients who have refractory solid tumors or hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose-limiting toxicity and maximum tolerated dose of perifosine administered as a varying series of loading and maintenance doses in patients with refractory solid tumors, non-Hodgkin's lymphoma, chronic lymphocytic leukemia, myelodysplastic syndromes, or Hodgkin's lymphoma.
* Determine the profile of adverse reactions (including changes in laboratory parameters) in patients treated with this regimen.
* Determine any disease responses that may occur in patients treated with this regimen.
* Determine the steady-state pharmacology and pharmacokinetics of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive a loading dose of oral perifosine on day 1 followed by a maintenance dose 2-3 times daily beginning on day 2 or 3 and continuing until day 21. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating loading and maintenance doses of perifosine until the maximum tolerated dose (MTD) of each is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional 10 patients are treated at that dose level.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A maximum of 45 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor, non-Hodgkin's lymphoma, chronic lymphocytic leukemia, myelodysplastic syndromes, or Hodgkin's lymphoma that has no effective standard therapeutic option but requires systemic therapy
* No history of CNS neoplasms
* For prostate cancer:

  * Tumor progression during blockade of testicular and adrenal androgens
  * At least 4 weeks since prior flutamide or other antiandrogens without disease improvement
  * Leuprolide or other gonadotropin-releasing hormones should be maintained in patients without an orchiectomy
  * Testosterone in the castrate range
* For breast cancer:

  * At least 4 weeks since any prior hormonal therapy with evidence of disease progression

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count greater than 50,000/mm^3
* Absolute granulocyte count greater than 500/mm^3
* Hemoglobin at least 9.0 g/dL

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT and SGPT no greater than 2.5 times normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No history of unstable or newly diagnosed angina pectoris
* No myocardial infarction within the past 6 months
* No New York Heart Association class II-IV heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No recent acute or chronic gastrointestinal conditions (e.g., stomach ulcer or enteritis) that might affect tolerability or drug absorption
* No allergic reaction to any medication with a structure similar to perifosine
* No pre-existing retinal disease or pathologic baseline electrooculogram
* No cataracts that would interfere with normal vision or require medical intervention
* No other serious concurrent illness that would preclude assessment of drug effect

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* At least 2 months since prior UCN-01
* More than 3 months since prior suramin

Endocrine therapy:

* See Disease Characteristics
* No concurrent corticosteroids except for physiological replacement or as antiemetics

Radiotherapy:

* At least 4 weeks since prior radiotherapy (6 weeks for bone-seeking radioisotopes) and recovered

Surgery:

* See Disease Characteristics

Other:

* No other concurrent antineoplastic therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08

CONTACTS AND LOCATIONS:
Overall Officials: Edward A. Sausville, MD, PhD, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland

REFERENCES:
- [Result] Monga M, Messmann RA, Headlee D, et al.: A phase I trial of oral perifosine in patients with refractory neoplasms. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1837, 7b, 2002.
- [Result] Messmann RA, Headlee D, Woo EW, et al.: A phase I trial of oral perifosine with different loading and maintenance schedules in patients with refractory neoplasms. [Abstract] Proc Am Assoc Cancer Res 42: A-2880, 2001.